CLINICAL TRIAL: NCT03281200
Title: A Multicentre, Retrospective Chart Review Study to Describe the Clinical Profile of Idiopathic Pulmonary Fibrosis (IPF) Patients Treated With Nintedanib (OFEV®) in Real-world Practice in Spain.
Brief Title: Chart Review Study to Describe the Clinical Profile of Idiopathic Pulmonary Fibrosis (IPF) Patients Treated With Nintedanib (OFEV®) in Real-world Practice in Spain
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0295
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Immunomodulating Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anatomical main group:
  Interventions: Drug: L - Antineoplastic and immunomodulating agents
- Therapeutic subgroup
  Interventions: Drug: L01 - Antineoplastic agents
- Pharmacological subgroup
  Interventions: Drug: L01X - Other antineoplastic agents
- Chemical subgroup
  Interventions: Drug: L01XE - Protein kinase inhibitors
- Chemical substance
  Interventions: Drug: L01XE31 - Nintedanib

INTERVENTIONS:
Drug: L - Antineoplastic and immunomodulating agents — L - Antineoplastic and immunomodulating agents
  Groups: Anatomical main group:
Drug: L01 - Antineoplastic agents — L01 - Antineoplastic agents
  Groups: Therapeutic subgroup
Drug: L01X - Other antineoplastic agents — L01X - Other antineoplastic agents
  Groups: Pharmacological subgroup
Drug: L01XE - Protein kinase inhibitors — L01XE - Protein kinase inhibitors
  Groups: Chemical subgroup
Drug: L01XE31 - Nintedanib — L01XE31 - Nintedanib
  Other Names: OVEF
  Groups: Chemical substance

SUMMARY:
The present study has been designed to characterize IPF patients treated with nintedanib (OFEV®), at time of treatment initiation, with respect to their clinical profile based on real-world data from January 2016 in Spanish Pulmonology Services.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years old
* The patient has IPF diagnosis according to most recent ATS/ERS/JRS/ALAT IPF guideline for diagnosis and management [5]
* The patient newly initiated treatment with nintedanib (OFEV®) since 01 January 2016 up to end of data collection date, according to the approved local Summary of Product Characteristics (SmPC)

Exclusion Criteria:

- Patients treated with nintedanib within a clinical trial or named-patient program or with any prior treatment of nintedanib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 175 IPF patients from 35 Pulmonology Services in Spain are planned to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dynamic solutions, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional study based on medical charts was conducted in approximately 35 pulmonology services in Spanish hospitals. Idiopathic pulmonary fibrosis (IPF) patients were characterized at the time of nintedanib initiation. Analysis of this report was performed using the data collected in the database from 21October2017 up to 31January2018.
Pre-assignment Details: All participants were screened for eligibility to participate in the study. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be analyzed if any one of the specific entry criteria were not met.
Groups:
- Total Patients With IPF: The IPF patients who initiated treatment with nintedanib (OFEV®) from 01January2016 up to 07June2018.
Period: Overall Study
Arm/Group | Total Patients With IPF
Started (Started are the treated with entry criteria met) | 172
Completed | 172
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients who met the selection criteria.
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of baseline visit
  Years | 71.0 (8.1)
Sex/Gender, Customized [Number; unit: Particpants]
  Male | 131
  Female | 40
  No data | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data was not collected for this trial.
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 170
  Asiatic | 1
  Arab | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Across Different Lung Function Categories (% FVC (Forced Vital Capacity))
Description: The distribution of patients across different lung function categories (% FVC serving as surrogate markers for IPF severity) of IPF patients treated with nintedanib (OFEV®) in routine clinical practice, at the time of treatment initiation.
Time Frame: From start of drug administration (01Jan16) until data collected in the database cut off date (31Jan18), i.e. Up to 765 days.
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentage of Patients (%)
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentage of Patients (%)
  Mild IPF: FVC ≥ 70% | 57.0
  Moderate IPF: FVC between 50% and 69% | 38.4
  Severe IPF: FVC < 50% | 4.7

2. Primary Outcome: Percentage of Patients Across Different Lung Function Categories (% DLCO (Diffusing Capacity of the Lungs for Carbon Monoxide))
Description: The distribution of patients across different lung function categories (% DLCO serving as surrogate markers for IPF severity) of IPF patients treated with nintedanib (OFEV®) in routine clinical practice, at the time of treatment initiation.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.Include only those patients DLCO value who has been answered in the case report form (CRF).
Measure: Number; unit: Percentage of Patients (%)
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 153
Percentage of Patients (%)
  Mild IPF: DLCO ≥ 50% | 42.5
  Moderate IPF: DLCO between 35% and 49% | 35.3
  Severe IPF: DLCO < 35% | 22.2

3. Secondary Outcome: The Demographic Baseline Characteristics - Age at the Time of Treatment Initiation
Description: The age of IPF patients at the time of treatment initiation with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Years | 70.1 (8.1)

4. Secondary Outcome: The Clinical Baseline Characteristics - Duration of the Disease
Description: Duration of the disease of IPF patients, calculated as the time elapsed from the date of diagnosis until the start date of treatment with OFEV® (years).
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Years | 1.5 (3.8)

5. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With Emphysema
Description: The percentage of patients with emphysema at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  No | 84.3
  Yes | 15.7

6. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With Usual Interstitial Pneumonia (UIP) Histopathological Pattern
Description: The usual interstitial pneumonia (UIP) histopathological pattern of IPF patients at the time of treatment initiation with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  No | 13.4
  Yes | 30.8
  No data | 55.8

7. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With UIP Radiological Pattern
Description: The UIP radiological pattern of IPF patients at the time of treatment initiation with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  No | 9.9
  Yes | 89.0
  No data | 1.2

8. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With the Initial Dose of OFEV®
Description: The percentage of patients initiated OFEV® dose of 150 milligram (mg)/ 12 hours (h) and 100 mg/12 h is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  150 mg/12 h | 88.4
  100 mg/12 h | 11.0
  No data | 0.6

9. Secondary Outcome: The Demographic Baseline Characteristics - Weight at the Start of Nintedanib Therapy
Description: The weight of IPF patients at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 160
Kilogram (Kg) | 77.1 (13.2)

10. Secondary Outcome: The Demographic Baseline Characteristics - Height at the Start of Nintedanib Therapy
Description: The height of IPF patients at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 159
Centimeters (cm) | 164.5 (8.9)

11. Secondary Outcome: The Demographic Baseline Characteristics - Body Mass Index (BMI) at the Start of Nintedanib Therapy
Description: The body mass index (BMI) of IPF patients at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Mean (Standard Deviation); unit: Kilogram/ meter^2 (kg/m^2)
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 159
Kilogram/ meter^2 (kg/m^2) | 28.4 (3.8)

12. Secondary Outcome: The Demographic Baseline Characteristics - 6-minute Walk Test
Description: The 6-minute walk test of IPF patients at the time of treatment initiation with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Mean (Standard Deviation); unit: Meter (m)
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 136
Meter (m) | 421.7 (118.6)

13. Secondary Outcome: The Demographic Baseline Characteristics - Percentage of Patients With Smoking Habit
Description: The percentage of patients with smoking habit at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentage of Participants
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentage of Participants
  Never smoker | 33.1
  Former smoker | 64.0
  Active smoker | 2.9

14. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With Dyspnoea
Description: The percentage of patients with dyspnoea at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Partients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Partients
  No | 5.2
  Yes | 93.0
  No data | 1.7

15. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With Exacerbations
Description: The percentage of patients with exacerbations of IPF in the year prior to initiating treatment is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of patients
  No | 84.9
  Yes | 11.6
  No data | 3.5

16. Secondary Outcome: The Clinical Baseline Characteristics - Percentage of Patients With Concomitant Treatments
Description: The percentage of patients taking any concomitant medication at the start of nintedanib therapy is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  No | 20.3
  Yes | 79.7

17. Secondary Outcome: Percentage of Patients With Prevalence of Comorbidity (Concomitant Diseases) at the Time of Treatment Initiation.
Description: The percentage of patients with comorbidity (concomitant diseases) at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  Hypertension | 45.9
  Dyslipidaemia | 42.4
  Gastroesophageal reflux | 25.6
  Diabetes mellitus | 19.8
  Emphysema | 15.7
  Cardiovascular disease | 15.7
  Obstructive sleep apnoea | 11.6
  Pulmonary hypertension | 5.8
  Lung cancer | 1.7
  Pulmonary infection | 1.2

18. Secondary Outcome: Percentage of Patients With Other Concomitant Diseases at the Time of Treatment Initiation.
Description: The percentage of patients with other concomitant diseases at the start of treatment with nintedanib (OFEV®) is presented.
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients | 41.9

19. Secondary Outcome: Percentage of Patients Distributed Across Different Lung Function Categories Based on the Reimbursement Threshold (%FVC)
Description: The distribution of patients across different lung function categories based on the reimbursement threshold (FVC >80%, 50-80%, and <50%).
Time Frame: as for outcome 1
Population: All enrolled patients who met the selection criteria.
Measure: Number; unit: Percentages of Patients
Arm/Group | Total Patients With IPF
Number analyzed (Participants) | 172
Percentages of Patients
  Mild IPF: FVC > 80% | 33.1 [26.3 to 40.8]
  Moderate IPF: FVC between 50% and 80% | 62.2 [54.5 to 69.4]
  Severe IPF: FVC < 50% | 4.7 [2.2 to 9.3]

ADVERSE EVENTS:
Time Frame: From start of drug administration (01Jan16) until final data set (07Jun18). i.e. Up to 889 days
Description: Patients who enrolled in the study and met the selection criteria used for reporting adverse events
Arm/Group | Total Patients With IPF
All-Cause Mortality (participants affected / at risk) | 10/172
Serious Adverse Events (participants affected / at risk) | 13/172
Other Adverse Events (participants affected / at risk) | 38/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Patients With IPF (N=172)
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Weight decreased (Investigations) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Patients With IPF (N=172)
Diarrhoea (Gastrointestinal disorders) | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03281200/Prot_SAP_000.pdf